CLINICAL TRIAL: NCT06655337
Title: Efficiency of the "Medidux" Smartphone App for Demission Management in Patients Medicated in Acute Admission Unit (AAU): a Randomized Controlled Trial.
Brief Title: Efficiency of the "Medidux" Smartphone App for Demission Management in Patients Medicated in Acute Admission Unit (AAU)
Acronym: EffiDux
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mobile Health AG (Industry)
Collaborators: Palleos Healthcare GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAUEffidux
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Acute Disease; Acute Hospitalization; Coughing; Back Pain; Abdominal Pain (AP); Patient Discharge; Patient Readmission; Mobile Health Apps; Mobile Health Technology (mHealth); Patient Reported Outcome (PRO)
Keywords: Acute Disease; Patient Discharge; Patient Readmission; Coughing; Back Pain; Abdominal Pain; Mobile Health Applications; Remote Monitoring; Post-discharge Care; Symptom Monitoring; Health Behaviour; Telemedicine; Randomized Controlled Trial
MeSH Terms: conditions — Acute Disease; Cough; Back Pain; Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: medidux App (Experimental): Participants in this arm will use the medidux™ smartphone application to monitor their symptoms and vital signs for 7 days following discharge from the Acute Admission Unit (AAU). The app provides health monitoring features, prompts for symptom tracking, and guidance on whether further medical consultation is required. Participants will log daily health data and receive automated reminders. The app aims to reduce post-discharge readmissions and emergency hospitalizations by providing real-time support. Follow-up assessments will be conducted at day 7 and day 28 post-discharge to evaluate symptom progression and healthcare utilization.
  Interventions: Device: Smartphone Application for Post-Discharge Symptom Monitoring
- Control Arm: Standard Post-Discharge Care (No Intervention): Participants in this arm will receive standard post-discharge care as currently practiced in the Acute Admission Unit (AAU). This may include follow-up calls or appointments with healthcare providers to monitor symptoms and progression after discharge, but participants will not use the medidux™ app for symptom tracking or monitoring. Follow-up assessments will be conducted at day 7 and day 28 post-discharge to evaluate symptom progression and healthcare utilization.

INTERVENTIONS:
Device: Smartphone Application for Post-Discharge Symptom Monitoring — This intervention involves the use of a smartphone application designed for symptom monitoring. The app enables participants to log daily health data, including symptoms and vital signs, for 7 days following discharge. It provides automated prompts and guidance for self-management, including when to seek medical assistance. The app does not provide direct medical intervention but facilitates remote symptom tracking to reduce readmissions and emergency hospitalizations. Follow-up consultations are conducted at day 7 and day 28.
  Arms: Intervention Arm: medidux App

SUMMARY:
The goal of this clinical trial is to evaluate whether the use of the medidux™ smartphone app can optimize post-discharge management for patients admitted to Acute Admission Units (AAU) with non-urgent health complaints. This trial includes adult patients (age ≥ 18) in Emergency Severity Index (ESI) triage system groups 4 (standard) or 5 (non-urgent), presenting with primary symptoms such as cough, back pain, or abdominal discomfort.

The main question it aims to answer is:

Can the medidux™ app reduce the incidence of AAU readmissions, emergency hospitalizations, or consultations with other medical providers within 7 days after initial admission?

Researchers will compare participants using the medidux™ app (intervention arm) with those receiving standard care (control arm) to observe potential differences in the rates of readmissions, emergency hospitalizations, and medical consultations.

Participants will:

* use the medidux™ app to monitor their symptoms and vital parameters for 7 days after discharge (intervention arm).
* receive follow-up consultations at day 7 and at day 28 to assess symptom progression and any healthcare interactions (both arms).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF)
* Age ≥ 18 years
* (Self-)admission to the involved Acute Admissions Unit (AAU)
* "Lead symptom" identified as coughing, back pain or abdominal discomfort
* Participant within ESI triage system group 4 (standard) and 5 (non-urgent)
* German-speaking
* Ownership of a smartphone or other mobile device with iOS or Android operating system

Exclusion Criteria:

* Age < 18 years
* Participant whose compliance to the study's protocol, e.g. due to mental health problems, physical problems, or the private life situation, can be justifiably doubted
* Participant with insufficient knowledge about the use of a smartphone or other mobile device with iOS or Android operating system
* Participant already using or planning to use another comparable electronic patient-reported symptom monitoring system (e.g. CANKADO) during this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Estimated)
Dates: Start 2025-09-28 (Actual); Primary Completion 2027-03-28 (Estimated); Study Completion 2027-03-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of AAU Readmissions, Emergency Hospitalizations, and Consultations of Other Medical Providers within 7 (± 1) days | 7 (± 1) days after the initial AAU admission
  This measure evaluates the number of participants who experience at least one AAU readmission, emergency hospitalization, or consultation with other medical providers within 7 days of the initial AAU admission. This is a binary measure (yes/no) indicating whether such an event has occurred.

SECONDARY OUTCOMES:
Incidence of AAU Readmissions, Emergency Hospitalizations, and Consultations of Other Medical Providers within 28 (± 1) days. | 28 (± 1) days after the initial AAU admission
  This measure captures the number of participants who experience at least one AAU readmission, emergency hospitalization, or consultation with other medical providers within 28 days of the initial AAU admission. This is a binary measure.
Incidence of AAU Readmissions within 7 (± 1) days | 7 (± 1) days after the initial AAU admission
  The number of participants who experience at least one readmission to the AAU within 7 days of their initial admission. This measure is a binary variable indicating whether a readmission has occurred.
Incidence of AAU Readmissions within 28 (± 1) days | 28 (± 1) days after the initial AAU admission
  The number of participants who experience at least one readmission to the AAU within 28 days of their initial admission. This is a binary variable indicating whether a readmission occurred.
Incidence of Emergency Hospitalizations within 7 (± 1) days | 7 (± 1) days after the initial AAU admission
  The number of participants who experience at least one emergency hospitalization within 7 days of their initial AAU admission. This is a binary variable indicating whether such an event occurred.
Incidence of Emergency Hospitalizations within 28 (± 1) days | 28 (± 1) days after the initial AAU admission
  The number of participants who experience at least one emergency hospitalization within 28 days of their initial AAU admission. This measure is a binary variable.
Incidence of Consultations of Other Medical Providers within 7 (± 1) days | 7 (± 1) days after the initial AAU admission
  This measure tracks the number of participants who consult with medical providers (outside of AAU or emergency hospitalizations) within 7 days of their initial AAU admission. It is a binary measure.
Incidence of Consultations of Other Medical Providers within 28 (± 1) days | 28 (± 1) days after the initial AAU admission
  This measure captures the number of participants who consult with medical providers within 28 days after their initial AAU admission. This is a binary variable.
Agreement Between ePRO-Derived AE Severity Index and Physician-Assessed AE Severity | 7 (± 1) days after the initial AAU admission
  This outcome assesses the agreement between the participant-reported ePRO-derived AE severity index (where 0.1 represents the least severe symptoms and 10 represents the most severe) and the AE severity index assessed by the investigator for one randomly selected symptom. The investigator uses a similar scale ranging from 0 (no symptoms) to 4 (severe symptoms). Agreement between the two assessments is calculated as a correlation coefficient.
Differences Between ePRO-Derived AE Severity and Physician-Assessed AE Severity Ratings | 7 (± 1) days after the initial AAU admission
  This outcome compares the differences between the participant-reported ePRO-derived AE severity index (ranging from 0.1 to 10, where higher scores represent more severe symptoms) and the investigator-assessed AE severity index (where 0 is no symptoms and 4 is severe symptoms) for a randomly selected symptom. The differences are presented in a cross-frequency table, showing any significant divergence between participant and physician assessments.
Number of Participant-Reported Symptoms by Severity | Daily over the 7 (± 1) day observation period
  This outcome counts the number of participant-reported symptoms as assessed through the ePRO-derived AE severity index, which ranges from 0.1 (least severe) to 10 (most severe). Scores are linearly transformed into an index from 0 to 4, where 0 represents no symptoms and 4 represents severe symptoms.
Evolution of Participant-Reported Symptoms Over Time | Daily over the 7 (± 1) day observation period
  This outcome tracks the progression of participant-reported lead symptoms over time, using the ePRO-derived AE severity index (0.1 to 10 scale, where 0.1 indicates least severity and 10 indicates most severity). The symptoms are reported daily, and the index is transformed linearly into an index from 0 (no symptoms) to 4 (severe symptoms).
Participant-Assessed Usability and Usefulness of the Smartphone App | Day 7 (± 1) after the initial AAU admission
  Usability and usefulness of the app will be assessed based on participant responses to an 11-point Likert scale questionnaire. Participants will rate usability and usefulness across several domains, with scores ranging from 0 (does not apply) to 10 (fully applies), where 0 represents the worst outcome and 10 represents the best possible outcome for each item, such as ease of use, helpfulness in symptom management, and perceived impact on physician consultations.

CONTACTS AND LOCATIONS:
Locations (1):
- Notfallzentrum See-Spital Horgen, Horgen, Canton of Zurich, Switzerland